CLINICAL TRIAL: NCT05681247
Title: Study on the Bioavailability and Bioequivalence of Ezetimibe Tablets in Healthy Subjects
Brief Title: Bioavailability and Bioequivalence of Ezetimibe Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SHX-BE-201703
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Hyperlipidemias
Keywords: Ezetimibe Tablet, Bioequivalence, Pharmacokinetics
MeSH Terms: conditions — Hyperlipidemias | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ezetimibe tablet (Experimental): ezetimibe tablet test formulation at a single dose of 10 mg
  Interventions: Drug: ezetimibe tablet
- ezetimibe tablet(Ezetrol ®) (Active Comparator): ezetimibe tablet reference formulation at a single dose of 10 mg
  Interventions: Drug: ezetimibe tablet(Ezetrol ®)

INTERVENTIONS:
Drug: ezetimibe tablet — The subjects randomly received single oral administration of ezetimibe tablet 10 mg
  Arms: ezetimibe tablet
Drug: ezetimibe tablet(Ezetrol ®) — The subjects randomly received single oral administration of ezetimibe tablet (Ezetrol ®) 10 mg.
  Arms: ezetimibe tablet(Ezetrol ®)

SUMMARY:
This study was conducted to assess the bioequivalence of the ezetimibe tablet to Ezetrol ® in healthy Chinese volunteers and estimate the pharmacokinetic proﬁles of ezetimibe tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects ≥18 years of age
* The body mass index is in the range of 18.0-26.0 kg/m2 (including the critical value).
* The weight of male is not less than 50.0 kg, and that of female is not less than 45.0 kg.
* Serum total cholesterol was between 2.9 and 5.0mmol/L (not including critical value).

Exclusion Criteria:

* any medical history of cardiovascular, digestive, respiratory, nervous or ematological diseases
* hepatic/renal impairment
* abnormal vital signs
* drug or alcohol abuse
* smoking ≥5 cigarettes per day ,
* donation(≥300ml) o
* enrollment in other clinical trials during the 3 months prior to screening
* allergic to ezetimibe or its excipients
* any use of other prescription drugs or vitamins or caffeine/xanthine-rich beverages 48h prior to taking medication
* lactating or pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-12-17 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) Peak Plasma Concentration (Cmax) | 80 days
  Peak Plasma Concentration (Cmax) Evaluation of Peak Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC)0-t | 80 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun F, Liu Y, Li T, Lin P, Jiang X, Li X, Wang C, Gao X, Ma Y, Fu Y, Cao Y. Pharmacokinetics and bioequivalence of Ezetimibe tablet versus Ezetrol(R):an open-label, randomized, two-sequence crossover study in healthy Chinese subjects. BMC Pharmacol Toxicol. 2023 Feb 3;24(1):7. doi: 10.1186/s40360-023-00649-y. PMID 36737825